CLINICAL TRIAL: NCT05520281
Title: ORPHYS - Short-term Psychodynamic Psychotherapy in Serious Physical Illness
Brief Title: Short-term Psychodynamic Psychotherapy in Serious Physical Illness
Acronym: ORPHYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKH70113404-2
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Malignant Neoplasm; Carcinoma; Palliative Care
Keywords: Advanced Cancer; Death anxiety; Demoralization; Existential distress; Mental disorders
MeSH Terms: conditions — Neoplasms; Carcinoma; Necrophobia; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Pre-Post Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Adult patients across all phases of advanced disease (UICC stage IV solid tumor) from diagnosis to terminal stages
  Interventions: Behavioral: Short-term psychodynamic psychotherapy for patients with serious physical illness (ORPHYS)

INTERVENTIONS:
Behavioral: Short-term psychodynamic psychotherapy for patients with serious physical illness (ORPHYS) — A short-term psychodynamic therapy that focuses on the special inner and outer situation of patients with a serious physical illness, especially with regard to the importance of relationships in a limited lifetime.

SUMMARY:
Life-threatening physical illness may powerfully re-activate existential conflict. There is little evidence to date on the effectiveness of relationship-focused therapies in this patient group.The aim of this study is to pilot a psychodynamic treatment for patients with advanced cancer and high psychological distress.

DETAILED DESCRIPTION:
Severely physically ill patients may experience existential distress symptoms including helplessness, hopelessness, death anxiety, perceived burdensomeness and a sense of pointlessness. The latter can significantly interfere with end-of-life care processes and outcomes (receipt of treatment according to preferences, expression of desire for hastened death). So far, empirically tested psychotherapeutic programs in advanced life-threatening illness have predominantly been ultra-short and applied supportive and resource-oriented techniques. Psychodynamic treatment allows to address clinically significant existential distress through its conceptualization from early relational life experiences.

The aim of this study is to pilot a psychodynamic treatment for patients with advanced cancer and high psychological distress.The inverstigators will

1. analyse the feasibility of the treatment, and
2. investigate changes in process- and patient-relevant outcomes over the course of the treatment

The inverstigators will conduct a single-group pre-post study with five assessment points in which 50 adult patients diagnosed with advanced cancer will receive a manualized psychodynamic short-term therapy. Target parameters are assessed by diagnostic interviews, focus interviews, self-assessment questionnaires as well as electronic patient records. For research objective b) the investigators will compare the intervention group with a matched comparison group of a longitudinal cohort sample (NCT04600206). Matching will be based on stress level, demographic, and medical parameters across the 5 assessment points.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* UICC stage IV solid tumor
* Informed consent
* Current physical condition that allows for at least 12 therapy sessions
* Indication: Presence of a mental disorder with existential stress and limitations in coping capacity

Exclusion Criteria:

* Acute suicidality
* Psychotic disorder (ICD-10: F2 diagnosis)
* Substance dependence or abuse (ICD-10: F1 diagnosis)
* Structural deficits that interfere with attending to regular appointments
* Other psychotherapeutic treatment
* Severe cognitive impairment
* Severe physical impairment
* Insufficient German to give informed consent and complete self-report questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | up to 12-months follow-up
  Will be assessed via Inventory for the Balanced Assessment of Negative Effects of Psychotherapy (INEP, Ladwig, Rief & Nestoriuc, 2014).
Acceptance | through study completion, an average of 6 months
  Will be assessed via drop-out rates (number of patients not completing at least 12 sessions) and treatment compliance (number of sessions missed).
Treatment adherence | through study completion, an average of 6 months
  Will be assessed via qualitative analysis of therapeutic session protocols and audio recordings.
Therapeutic competence | through study completion, an average of 6 months
  Will be assessed via qualitative analysis of supervision protocols.
Treatment feasibility | through study completion, an average of 6 months
  Will be assessed via semi-structured qualitative interviews.

SECONDARY OUTCOMES:
Therapeutic alliance I | 3-, 6- 9- and 12-months follow-up
  Will be assessed via California Psychotherapy Alliance Scales (CALPAS, Marmar & Gaston, 1989) for patients and therapists.
Interpersonal problems | Baseline, 3-, 6-, 9- and 12-months follow up
  Will be assessed via inventory for assessment of interpersonal problems (IIP-D-32, Thomas, Brähler & Strauß, 2011).
Therapeutic process | through study completion, an average of 6 months
  Will be assessed via semi-structured qualitative interviews.
Therapeutic alliance II | 3-, 6- 9- and 12-months follow-up
  Will be assessed via Helping Alliance Questionnaire (HAQ, Luborsky et al., 1996) (IIP-D-32, Thomas, Brähler & Strauß, 2011) for patients and therapists.

OTHER OUTCOMES:
Desire for hastened death | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the short form of the Schedule of Attitudes Toward Hastened Death (SAHD-A, Kolva et al., 2017).
Suicidal ideation | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the Beck Scale for Suicidal Ideation (BSS, Kliem & Brähler, 2015).
Coping and Demoralisation | a) Baseline and 6-months follow-up, b) Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the a) Structured Interview for Psychological Adjustment and Demoralisation (Bobevski & Kissane, 2019) and b) Demoralisation Scale-II (DS-II, Robinson et al., 2016).
Prevalence of adjustment disorder | Baseline and 6-months follow-up
  Will be assessed according to International Classification of Diseases (ICD-11) using the Adjustment Disorder Module of the CIDI (Composite International Diagnostic Interview, (Perkonigg et al., 2018).
Aggressiveness of care | 4 weeks prior to death
  Will be assessed according to the criteria by Earle et al., 2003: receipt of chemotherapy in the last two weeks of life, emergency hospital admissions or intensive-care treatment during the last month of life. Will be obtained from medical chart reviews for deceased patients.
Prevalence of affective and anxiety disorders | Baseline and 6-months follow-up
  Will be assessed using the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID-5, Beesdo-Baum et al., 2019).
Death Anxiety | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the Death Anxiety and Distress Scale (DADDS, Krause etal., 2015).
Perceived Relatedness | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using Subscales (Dependence, Relatedness) of the Depressive Experience Questionnaire (DEQ, Blatt, D'Afflitti & Quinlan, 1976; Blatt et al., 1982).
End-of-life preparation and adaption | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the Revised Loss Orientation and Life Engagement in Advanced Cancer Scale (LOLES, Vehling et al., 2018).
Dignity related distress | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the Sense of Dignity Item (SDI, Chochinov et al., 2002) and the Patient Dignity Inventory (PDI, Chochinov, 2008).
Meaningfulness in life and crisis of meaning | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the Sources of Meaning and Meaning in Life Questionnaire (SoMe, Schnell, 2009).
Quality of life at the end of life | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using a subscale (Life completion) of the Quality of Life at the End of Life-Cancer-Psychosocial Questionnaire (Qual-EC-P).
Coping resources | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using subscales (coping competence, adaptability) of the questionnaire for patient competence in coping with cancer (PCQ, Aderhold et al., 2019).
Need for and utilisation of psychosocial support for existential distress | Baseline, 3-, 6-, 9- and 12-months-follow-up
  Will be assessed using the Structured questionnaire of psychosocial support needs for existential distress.

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Vehling, PD, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (4):
- Germany (4):
  - Clinical Institute for Psychosomatic Medicine and Psychotherapy, University Medical Center Düsseldorf, Düsseldorf
  - University Medical Center Hamburg Eppendorf, Department of Medical Psychology, Hamburg
  - Institute of Social Work, University of Kassel, Kassel
  - Psychosomatics, Psychotherapy and Psychooncology, Medicine II, University of Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No